CLINICAL TRIAL: NCT05938530
Title: Sirolimus Drug-coated Balloon Versus Stent Graft for Thrombosed Arteriovenous Graft (SUSTAIN)
Brief Title: Sirolimus Drug-coated Balloon Versus Stent Graft
Acronym: SUSTAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOH-CNIG21nov-0008
Record Dates: First submitted 2023-06-26; First posted 2023-07-10 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Arteriovenous Shunt Thrombosis; Blood Vessel Prosthesis
Keywords: Arteriovenous graft; Thrombosis; Sirolimus; Drug-coated balloon; stent graft
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated in a 1:1 ratio into either the treatment (sirolimus DCB) arm or control (stent graft) arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sirolimus drug-coated balloon (Experimental): The trial product is MagicTouch sirolimus drug coated balloon (Concept Medical). Sirolimus will be transferred from the balloon to the graft vein junction by inflating the balloon for 2 minutes at rated burst pressure (typically 12 to 14ATM).
  Interventions: Device: Sirolimus drug-coated balloon
- Stent graft (Active Comparator): Stent graft is the current standard of care for treatment of arteriovenous graft malfunction. A stent graft will be deployed at the graft vein junction.
  Interventions: Device: Stent graft

INTERVENTIONS:
Device: Sirolimus drug-coated balloon — The effectiveness of sirolimus coated balloon in patients with dialysis access dysfunction has been shown in a small pilot study in the salvage of thrombosed arteriovenous graft.
  Arms: Sirolimus drug-coated balloon
Device: Stent graft — Stent graft has been shown to be superior than plain balloon angioplasty in the treatment of AVG dysfunction.
  Arms: Stent graft

SUMMARY:
A functioning dialysis vascular access is critical to the delivery of lifesaving hemodialysis. Arteriovenous graft (AVG) is a surgically created vascular access used for hemodialysis in patients with end-stage renal disease. AVG thrombosis due to underlying flow-limiting stenosis of the graft vein junction and outflow veins is a common complication. Thrombosed AVG can be treated with thrombolysis combined with percutaneous transluminal angioplasty with good immediate success rates. However, the mid-to-long term patency rates following angioplasty have been suboptimal. Sirolimus drug-coated balloon has been shown to be safe and effective in the salvage of thrombosed arteriovenous graft. The investigators hypothesize that sirolimus drug-coated balloon is non-inferior to stent graft in maintaining the patency of thrombosed AVG that is successfully salvaged. This study is conducted to compare the 6-month access circuit primary patency of thrombosed AVG treated with sirolimus drug-coated balloon versus stent graft.

DETAILED DESCRIPTION:
Arteriovenous graft (AVG) is a surgically created vascular access used for hemodialysis (HD). Neointimal hyperplasia frequently occurs within AVG, resulting in flow-limiting stenosis and thrombosis. The primary patency rates of AVGs after creation were 58% at 6 months and 33% at 18 months. Hence, vascular access failure has been a common reason for hospitalization among HD patients. The culprit lesion in AVG thrombosis is usually the graft-vein (GV) junction stenosis. Histopathology examination of thrombosed AVG demonstrated maximal neointimal hyperplasia at the GV junction. Thrombolysis combined with percutaneous transluminal angioplasty (PTA) of underlying stenosis has been the standard of care to restore the function of thrombosed AVGs. Despite its widespread availability and minimally invasive nature, the mid- and long-term patency of PTA for thrombosed AVG is far from satisfactory. The reported access circuit primary patency (ACPP) rate of thrombosed AVG following thrombolysis combined with PTA alone was only 23.5% at 6-month. This is because PTA is purely a mechanical intervention that does not address the underlying biological process of neointimal hyperplasia.

Stent graft is a type of vascular stent with expanded polytetrafluoroethylene (ePTFE) coating. It provides mechanical scaffolding that keeps vascular lumen open while the ePTFE coating limits neointimal hyperplasia. The therapeutic efficacy of stent graft in the treatment of graft vein junction stenosis has been convincingly demonstrated in several randomized controlled trials (RCTs). For thrombosed AVG, the reported access circuit primary patency rates at 6-month following stenting were 34% compared to 21.8% with PTA alone. The National Kidney Foundation Kidney Disease Outcomes Quality Initiative (KDOQI) Clinical Practice Guideline for Vascular Access: 2019 Update therefore suggests the use of stent-grafts in preference to PTA alone to treat clinically significant GV junction stenosis in AVG for a better 6-month postintervention outcome. Despite its superiority compared to PTA in maintaining the short- and long-term patency of thrombosed AVG, stent graft is expensive and may not be suitable for all patients as it could impede future surgical revision or creation of a secondary vascular access in the ipsilateral arm. Furthermore, the deployment of stent graft is technically challenging and requires refined interventional skills in experience hands to ensure accurate landing and prevent migration.

Drug-coated balloon (DCB) is a balloon catheter that is coated with an anti-proliferative drug. The drug is delivered directly to the vessel wall upon balloon inflation to prevent neointimal hyperplasia and restenosis. The efficacy of DCB have been shown in several randomized controlled trials. Liao et al demonstrated that angioplasty with DCB resulted in a modest improvement in primary patency of AVG with GV junction stenosis. We conducted a prior pilot study to examine the feasibility of Sirolimus DCB angioplasty at the GV junction following successful PTA for thrombosed AVGs. Our study demonstrated an ACPP of 55% at 6 months. This finding could imply that Sirolimus DCB can be an alternative option to stent graft deployment which is the recommended treatment. DCBs are cheaper and will not impede future secondary vascular access creation. Furthermore, DCB angioplasty is similar to PTA with plain balloon procedurally, thus it is not as technically challenging as stent graft deployment and does not require highly skilled operators.

The investigators aim to perform a single-centre 2-arm parallel randomized non-inferiority trial to compare the 6-month post-intervention access circuit primary patency (ACPP) of sirolimus DCB versus stent graft in the management of thrombosed AVG.

RECRUITMENT Patients who are admitted to the hospital for thrombosed AVG will be screened and offered enrollment if they meet the inclusion criteria. Patients will be consented if they fulfill the preliminary eligibility criteria and agree to participate in the study. Patients who have successful thrombectomy of the AVG is entered to the trial and randomized to receive either sirolimus DCB or stent graft. Patients who are unsuitable for the trial will be treated in the according to hospital standard protocol.

STUDY PROCEDURE Thrombolysis of the AVG will be performed as per standard hospital protocol. Briefly, an antegrade and retrograde vascular sheath will be placed in the thrombosed AVG under ultrasound guidance. Thrombolytic agents will be delivered into the thrombosed AVG via the vascular sheaths or catheters. The culprit venous stenosis will be treated using plain angioplasty balloon and thrombus within the AVG macerated using the same angioplasty balloon. If needed, the arterial plug will be dislodged by a 5.5Fr Fogarty balloon. Following successful thrombolysis of the AVG, the number and location of lesions within the dialysis circuit will be documented. After successful thrombolysis and adequate angioplasty of the GV junction (defined as <30% residual stenosis after treatment at rated burst pressure of the angioplasty balloon), patient will be randomized to either receive sirolimus DCB or stent graft deployment at the GV junction. To ensure adequate contact, the DCB or stent graft should be of the same or oversized by 1mm the diameter of the AVG. The DCB will be inflated up to the manufacturer's stated burst pressure. An inflation device with a pressure gauge will be used to inflate up to manufacturers' stated burst pressure for a duration of 2 minutes. For patients who are randomized to stent graft, a same diameter plain angioplasty balloon will be used to fully expand the stent graft after deployment. Post treatment with DCB or stent graft, a completion graftogram will be done to document the results. The size of the balloon/stent used, inflation pressure, number of inflations, procedure complications (if any), and residual stenosis will be recorded.

POST-PROCEDURE REVIEW AND FOLLOW-UP

Immediate Post-intervention Follow-up

All participants will be assessed by physical examination for the presence of a palpable, continuous thrill as a measure of technical success. Clinical success is defined as the patient's ability to undergo at least one hemodialysis treatment at the prescribed blood flow rate for the prescribed treatment duration.

Post-intervention 1-month Follow-up

All patients will be contacted via phone at 1-month ± 2 weeks to assess for any treatment site-related adverse event within 30 days.

Post-intervention 6-month Follow-up

The participant returns for a 6-month ± 4 weeks follow-up in the clinic to be assessed by the study team for the patency rate of AVG: a palpable, continuous thrill. Dialysis charts will be reviewed for clinical indicators of significant stenosis.

Post-intervention 12-month Follow-up

Each patient will be followed-up in clinic at 12-month ± 4 weeks follow-up in the clinic to be assessed by the study team for the patency rate of AVG: a palpable, continuous thrill. Dialysis charts will be reviewed for clinical indicators of significant stenosis.

Reintervention Participants who required repeat thrombolysis of the AVG are considered to have reached primary endpoint and deemed to have completed the study and will not be replaced. The study team will continue tracking their progress until the end of intended 12-month study participation. The tracking includes review of their medical records, and if necessary, telephone call to the patient, to complete the data collection.

Expected duration of study The total duration of study for each patient upon randomization will be 12-months. The study ends after the 12-month clinic follow-up.

*Patency definitions are defined based on SIR reporting standards (Gray et al., 2003):

Post-intervention target lesion patency:

Interval after intervention until the next re-intervention at graft vein junction or until the access is abandoned. Percutaneous or surgical treatments of a new arterial or venous outflow stenosis/occlusion (including access thrombosis) that do not involve or exclude the graft vein junction from the access circuit are compatible with lesion patency. The creation of new access that incorporates the graft vein junction into the new access circuit is also compatible with target lesion patency.

Post-intervention access circuit primary patency:

Interval following intervention until the next access thrombosis or repeated intervention. It ends with the treatment of a lesion anywhere within the access circuit, from the arterial inflow to the superior vena cava-right atrial junction.

Post-intervention access circuit assisted primary patency:

Interval after intervention until access thrombosis or surgical intervention that excludes the treated lesion from the access circuit. Percutaneous treatments of either restenosis/occlusion of the previously treated lesion or a new arterial or venous outflow stenosis/occlusion (excluding access thrombosis) are compatible with assisted primary patency.

Post-intervention access circuit secondary patency:

Interval after intervention until the access is surgically declotted, revised or abandoned. Thrombolysis and percutaneous thrombectomy are compatible with secondary patency.

^Complications will be categorized according to SIR definitions of minor or major complications (Aruny et al., 2003):

A major complication is defined as one that:

1. require therapy, minor hospitalization (< 48 hours),
2. require major therapy, unplanned increase in the level of care, prolonged hospitalization (>48 hours),
3. leads to permanent adverse sequelae, or
4. death

A minor complication is one that:

1. requires no therapy with no consequence,
2. requires nominal therapy with no consequence; includes overnight admission for observation only.

ELIGIBILITY:
Inclusion Criteria:

* Thrombosed AVG in the upper arm
* Successful thrombolysis of the thrombosed AVG, defined as the re-established of flow on Digital Subtraction Angiography (DSA) and restoration of thrill in the AVG on clinical examination (to be determined during procedure)

Exclusion Criteria:

* Patient unable to provide informed consent
* Previous bare metal stent or stent-graft placement within the dialysis access
* Previous treatment with DCB within 3 months
* Presence of central vein stenosis which cannot be adequately treated (residual recoil of more than 30%)
* Failure to re-establish blood flow
* Failure to adequately treat the GV junction (defined as residual stenosis of more than 30%)
* Sepsis or active infection
* Recent intracranial bleed or gastrointestinal bleed within the past 12 months
* Allergy to iodinated contrast media, anti-platelet drugs, heparin or sirolimus
* Pregnancy
* Life expectancy < 12 months based on physician's estimate (eg. active malignancy)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Access circuit primary patency of AVG at 6-months | 6 months
  This is measured by the percentage of patients whose AVG remain patent at 6 months after the procedure

SECONDARY OUTCOMES:
Access circuit primary patency of AVG at 12-months | 12 months
  This is measured by the percentage of patients whose AVG remain patent at 12 months after the procedure
Target lesion primary patency at 6- and 12-months | 6 and 12 months
  This is measured by the percentage of patients whose graft vein junction of AVG remain intervention-free at 6 and 12 months
The number of interventions needed to maintain patency of AVG at 12 months | 12 months
  Total number of repeat interventions to treat the AVG in 12 months
The technical and clinical success rates of the procedures | Immediately after the procedure
  The percentage of patients who have successful re-establishment of flow in AVG (technical success) and undergo hemodialysis at prescribed blood flow for the prescribed duration (clinical success)
The complication rates of the procedures | Immediately after the procedure
  Complication rates of the procedures
The cost associated with AVG interventions within 12 months | 12 months
  Total healthcare spending for AVG interventions

CONTACTS AND LOCATIONS:
Overall Officials: Ru Yu Tan, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 2021 USRDS Annual Data Report: Epidemiology of kidney disease in the United States. National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD.
- [Background] Singapore Renal Registry Annual Report 2019
- [Background] Roy-Chaudhury P, Kelly BS, Miller MA, Reaves A, Armstrong J, Nanayakkara N, Heffelfinger SC. Venous neointimal hyperplasia in polytetrafluoroethylene dialysis grafts. Kidney Int. 2001 Jun;59(6):2325-34. doi: 10.1046/j.1523-1755.2001.00750.x. PMID 11380837
- [Background] Huber TS, Carter JW, Carter RL, Seeger JM. Patency of autogenous and polytetrafluoroethylene upper extremity arteriovenous hemodialysis accesses: a systematic review. J Vasc Surg. 2003 Nov;38(5):1005-11. doi: 10.1016/s0741-5214(03)00426-9. PMID 14603208
- [Background] Lee T, Roy-Chaudhury P. Advances and new frontiers in the pathophysiology of venous neointimal hyperplasia and dialysis access stenosis. Adv Chronic Kidney Dis. 2009 Sep;16(5):329-38. doi: 10.1053/j.ackd.2009.06.009. PMID 19695501
- [Background] Vesely T, DaVanzo W, Behrend T, Dwyer A, Aruny J. Balloon angioplasty versus Viabahn stent graft for treatment of failing or thrombosed prosthetic hemodialysis grafts. J Vasc Surg. 2016 Nov;64(5):1400-1410.e1. doi: 10.1016/j.jvs.2016.04.035. Epub 2016 Jun 25. PMID 27353358
- [Background] Haskal ZJ, Trerotola S, Dolmatch B, Schuman E, Altman S, Mietling S, Berman S, McLennan G, Trimmer C, Ross J, Vesely T. Stent graft versus balloon angioplasty for failing dialysis-access grafts. N Engl J Med. 2010 Feb 11;362(6):494-503. doi: 10.1056/NEJMoa0902045. PMID 20147715
- [Background] Haskal ZJ, Saad TF, Hoggard JG, Cooper RI, Lipkowitz GS, Gerges A, Ross JR, Pflederer TA, Mietling SW. Prospective, Randomized, Concurrently-Controlled Study of a Stent Graft versus Balloon Angioplasty for Treatment of Arteriovenous Access Graft Stenosis: 2-Year Results of the RENOVA Study. J Vasc Interv Radiol. 2016 Aug;27(8):1105-1114.e3. doi: 10.1016/j.jvir.2016.05.019. Epub 2016 Jul 4. PMID 27388566
- [Background] Lok CE, Huber TS, Lee T, Shenoy S, Yevzlin AS, Abreo K, Allon M, Asif A, Astor BC, Glickman MH, Graham J, Moist LM, Rajan DK, Roberts C, Vachharajani TJ, Valentini RP; National Kidney Foundation. KDOQI Clinical Practice Guideline for Vascular Access: 2019 Update. Am J Kidney Dis. 2020 Apr;75(4 Suppl 2):S1-S164. doi: 10.1053/j.ajkd.2019.12.001. Epub 2020 Mar 12. PMID 32778223
- [Background] Kitrou PM, Katsanos K, Spiliopoulos S, Karnabatidis D, Siablis D. Drug-eluting versus plain balloon angioplasty for the treatment of failing dialysis access: final results and cost-effectiveness analysis from a prospective randomized controlled trial (NCT01174472). Eur J Radiol. 2015 Mar;84(3):418-423. doi: 10.1016/j.ejrad.2014.11.037. Epub 2014 Dec 15. PMID 25575743
- [Background] Irani FG, Teo TKB, Tay KH, Yin WH, Win HH, Gogna A, Patel A, Too CW, Chan SXJM, Lo RHG, Toh LHW, Chng SP, Choong HL, Tan BS. Hemodialysis Arteriovenous Fistula and Graft Stenoses: Randomized Trial Comparing Drug-eluting Balloon Angioplasty with Conventional Angioplasty. Radiology. 2018 Oct;289(1):238-247. doi: 10.1148/radiol.2018170806. Epub 2018 Jul 24. PMID 30040057
- [Background] Swinnen JJ, Hitos K, Kairaitis L, Gruenewald S, Larcos G, Farlow D, Huber D, Cassorla G, Leo C, Villalba LM, Allen R, Niknam F, Burgess D. Multicentre, randomised, blinded, control trial of drug-eluting balloon vs Sham in recurrent native dialysis fistula stenoses. J Vasc Access. 2019 May;20(3):260-269. doi: 10.1177/1129729818801556. Epub 2018 Sep 18. PMID 30227772
- [Background] Lookstein RA, Haruguchi H, Ouriel K, Weinberg I, Lei L, Cihlar S, Holden A; IN.PACT AV Access Investigators. Drug-Coated Balloons for Dysfunctional Dialysis Arteriovenous Fistulas. N Engl J Med. 2020 Aug 20;383(8):733-742. doi: 10.1056/NEJMoa1914617. PMID 32813949
- [Background] Liao MT, Lee CP, Lin TT, Jong CB, Chen TY, Lin L, Hsieh MY, Lin MS, Chie WC, Wu CC. A randomized controlled trial of drug-coated balloon angioplasty in venous anastomotic stenosis of dialysis arteriovenous grafts. J Vasc Surg. 2020 Jun;71(6):1994-2003. doi: 10.1016/j.jvs.2019.07.090. Epub 2019 Oct 11. PMID 31611105
- [Background] Tan CW, Tan RY, Pang SC, Tng ARK, Tang TY, Zhuang KD, Chua JME, Tay KH, Chong TT, Tan CS. Single-Center Prospective Pilot Study of Sirolimus Drug-Coated Balloon Angioplasty in Maintaining the Patency of Thrombosed Arteriovenous Graft. J Vasc Interv Radiol. 2021 Mar;32(3):369-375. doi: 10.1016/j.jvir.2020.11.010. Epub 2020 Dec 15. PMID 33334667